CLINICAL TRIAL: NCT00368550
Title: Sertraline Pharmacotherapy for Alcoholism Subtypes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Henry R. Kranzler, M.D., University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-225-2; R01AA013631 (NIH)
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Alcoholism
Keywords: Alcohol Drinking; Alcohol Dependence; Sertraline Pharmacotherapy; Alcoholism Subtypes; Early- versus Late-Onset Alcoholism
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral sertraline, cognitive-behavioral counseling to maintain abstinence from alcohol
  Interventions: Drug: Sertraline
- 2 (Placebo Comparator): Placebo, cognitive-behavioral counseling to maintain abstinence from alcohol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Sertraline (to a maximum of 200 mg/day) for 14-week treatment period
  Other Names: Zoloft
  Arms: 1
Drug: Placebo — Placebo for 14-week treatment period
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Sertraline, compared to placebo, is effective in the treatment of alcohol dependence as a function of the subtype of alcoholic patient being treated. This involved administering sertraline (to a maximum of 200 mg/day) or an inactive placebo for a 14-week treatment period.

DETAILED DESCRIPTION:
In an effort to broaden the options for pharmacotherapy of alcoholism, this study will examine the effects of sertraline, a selective serotonin reuptake inhibitor (SSRI), for the treatment of alcohol dependence. The study is based on evidence that, although SSRI therapy is not appropriate for all alcoholics, there exists a substantial subgroup of alcoholics for whom SSRIs appear to exert a clinically important effect. Sertraline is among the most widely prescribed psychotropic medications in the world. Consequently, this study will examine the safety and efficacy of sertraline, the mechanism and duration of those effects and the best method for subtyping alcoholics to identify individuals for whom the medication is most likely to produce a clinically important reduction in drinking behavior.

The study employs a parallel-group, prospective design in which randomization is balanced on patient subtype (early-onset/late-onset) and other relevant pretreatment measures with an approximately equal number of subjects assigned to treatment with sertraline (to a maximum of 200 mg/day) or placebo. The study will include a 14-week treatment period; because the 2 weeks are for medication taper, efficacy will be evaluated over the first 12 treatment weeks. A total of 160 early-onset or late-onset alcoholics will be randomized. Daily process measures of positive and negative events, global perceived stress, mood, desire to drink, and drinking frequency and intensity, collected using interactive voice response technology, will provide insight into the mechanisms by which sertraline may exert its effects. Coping-skills training will be provided weekly for the first 6 weeks, then every other week for the last 8 weeks of the study. A 6-month post-treatment follow-up period will evaluate the duration of medication effects. This study will also examine the relation between genotypes at a number of relevant loci and both risk of alcohol dependence and response to sertraline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current episode (i.e., in the preceding month) of alcohol dependence defined by Diagnostic and Statistical Manual of Mental Disorders 4th ed (DSM-IV) criteria
* 18-65 years of age
* Abstinent from alcohol for a period of at least 3 days prior to baseline research assessment
* Able to read English and complete study evaluations
* Male, or if female, without active reproductive potential
* Participants will have signed informed consent

Exclusion Criteria:

* Currently meets criteria for dependence on a psychoactive substance other than alcohol and nicotine
* Regular use of psychoactive drugs including anxiolytics and antidepressants
* Current use of disulfiram or naltrexone
* Current major depression or psychosis (or other severe psychiatric disability e.g., suicidality, current mania)
* Significant underlying medical conditions such as hepatic, cerebral, renal, thyroid, or cardiac pathology, which in the opinion of the evaluating physician would preclude the patient from study adherence or be of potential harm to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R. Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Kranzler HR, Armeli S, Tennen H, Covault J. 5-HTTLPR genotype and daily negative mood moderate the effects of sertraline on drinking intensity. Addict Biol. 2013 Nov;18(6):1024-31. doi: 10.1111/adb.12007. Epub 2012 Nov 12. PMID 23145795
- [Derived] Kranzler HR, Armeli S, Tennen H. Post-treatment outcomes in a double-blind, randomized trial of sertraline for alcohol dependence. Alcohol Clin Exp Res. 2012 Apr;36(4):739-44. doi: 10.1111/j.1530-0277.2011.01659.x. Epub 2011 Oct 7. PMID 21981418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from Feb. 2004 to March 2009 through advertisements and referrals by area clinicians.
Pre-assignment Details: All patients underwent physical examination and routine laboratory testing during screening. 143 prospective patients were screened, of which 4 did not meet study criteria and 5 chose not to participate.
Groups:
- Sertraline: Sertraline plus coping skills therapy. Medication to a maximum of 200 mg/day orally in two doses. Coping skills therapy, aimed at improving patients' ability to change their drinking behavior, was provided at each visit.
- Placebo: Placebo plus coping skills therapy. Coping skills therapy, aimed at improving patients' ability to change their drinking behavior, was provided at each visit.
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 63 | 71
Completed | 35 | 48
Not Completed | 28 | 23
Not completed — Adverse Event | 7 | 4
Not completed — Lack of Efficacy | 4 | 9
Not completed — Withdrawal by Subject | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 63 | 71 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 71 | 133
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.1) | 47.3 (9.5) | 47.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 51 | 57 | 108
Region of Enrollment [Number; unit: participants]
  United States | 63 | 71 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Days on Which Subjects Drank
Description: Obtained using daily interactive voice response data augmented by Timeline Followback data. Missing days were treated as drinking days.
Time Frame: 12-week treatment period
Population: All randomized subjects with missing days imputed as drinking days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 63 | 71
days | 37.0 (30.6) | 33.8 (27.3)

2. Secondary Outcome: Number of Days of Heavy Drinking (Defined as Days on Which Women Drank >= 4 Drinks and Men Drank >= 5 Drinks)
Description: Obtained using daily interactive voice response data augmented by Timeline Followback data. Missing days were treated as heavy drinking days.
Time Frame: 12-week treatment period
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 63 | 71
days | 31.9 (29.0) | 26.4 (26.4)

3. Secondary Outcome: Change in the Level of Alcohol-related Problems
Description: Measured using the SIP (Short Inventory of Problems), which was administered at pretreatment and at the end of treatment. The range of scores on the SIP is 0 (no alcohol-related problems) to 45 (most severe alcohol-related problems) and the time frame for reporting is the preceding 3 months. The data presented here represent a difference score of treatment minus baseline.
Time Frame: 12-week treatment period compared with baseline value
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 63 | 71
Units on a scale | 6.0 (9.2) | 9.0 (9.5)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Items used to monitor the occurrence of adverse events are those identified in previously completed efficacy studies of sertraline.
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 3/63 | 0/71
Other Adverse Events (participants affected / at risk) | 22/63 | 14/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=63) | Placebo (N=71)
Hospitalization due to chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization due to relapse to heavy drinking (Psychiatric disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=63) | Placebo (N=71)
agitation (Psychiatric disorders) | 2 (2) | 5 (5)
nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
insomnia (Psychiatric disorders) | 6 (6) | 7 (8)
diarrhea (Gastrointestinal disorders) | 16 (21) | 10 (13)
sexual problems (Reproductive system and breast disorders) | 15 (17) | 3 (4)
tired/sleepy (Nervous system disorders) | 13 (15) | 4 (4)
decreased appetite (Nervous system disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No